CLINICAL TRIAL: NCT05546086
Title: Risk Prediction System for Metabolic Associated Fatty Liver Disease, a Community-based Cohort Study
Brief Title: BeijngFH Health Cohort Study
Acronym: FHCS
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: CFH2022-1-2021
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Non-Alcoholic Fatty Liver Disease; Cohort Studies; Risk Factors
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Metabolic associated fatty liver disease(MEFLD) is a major chronic liver disease that can lead to various adverse events, such as liver cancer, cardiovascular disease, and chronic kidney disease. The present community-based cohort study enrolls subjects who take health physical examinations at the sub-center outpatient department, Beijing Friendship Hospital. Investigators collect their baseline information, including demographic data, clinical history, physical examination, laboratory results, imageological examination, and so on. Follow-up surveys are conducted annually and the information collected is the same as the baseline. The outcome information, including cardiovascular disease, malignancy, liver cirrhosis, liver decompensation, liver transplantation, and all-cause mortality, are obtained by linking to the hospital discharge database and death registration system of Beijing. The primary aim of the study is to build a risk-stratified evaluation system for MAFLD through the cohort.

DETAILED DESCRIPTION:
The present community-based cohort study enrolls subjects who take physical health examinations at the sub-center outpatient department, Beijing Friendship Hospital. After signing the informed consent, Their previous health physical examination results, which were recorded in the Hospital Information System (HIS) are collected retrospectively. Then, Investigators collect their baseline information, including demographic data, clinical history, physical examination, laboratory results, image logical examination, and so on. Additionally, follow-up surveys will be conducted annually and the information collected is the same as the baseline. The outcome information, including cardiovascular disease, malignancy, liver cirrhosis, liver decompensation, liver transplantation, and all-cause mortality, is obtained from the hospital discharge database and death registration system in Beijing. The study's primary aim is to build a risk-stratified evaluation system for MAFLD through a community population cohort with long-term stable follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Permanent residents in Beijing
* Signing informed consent

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The present community-based cohort study enrolls subjects who take health physical examinations at the sub-center outpatient department, Beijing Friendship Hospital from April 2022.
Sampling Method: Non-Probability Sample
Enrollment: 8103 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2032-04-18 (Estimated); Study Completion 2032-04-18 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular disease | 1 to 10 years
  Incidence of cardiovascular disease during follow-ups

SECONDARY OUTCOMES:
Malignancy | 1 to 10 years
  Incidence of malignancy during follow-ups
Liver cirrhosis | 1 to 10 years
  Incidence of liver cirrhosis during follow-ups
Liver decompensation | 1 to 10 years
  Incidence of liver decompensation during follow-ups
Liver transplantation | 1 to 10 years
  Incidence of liver transplantation during follow-ups
All-cause mortality | 1 to 10 years
  Incidence of all-cause mortality during follow-ups

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No